CLINICAL TRIAL: NCT05315908
Title: COVID-19 Testing in Underserved and Vulnerable Populations Receiving Care in San Diego Community Health Centers
Brief Title: COVID-19 Testing in Underserved and Vulnerable Populations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of low testing uptake, slow accrual at participating health centers and continuously changing COVID pandemic, research investigators had to terminate the original study and consider alternate strategies.
Sponsor: Jesse Nodora (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jesse Nodora, Assoc Adjt Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201505; 3UH3CA233314-02S1 (NIH)
Record Dates: First submitted 2022-01-22; First posted 2022-04-07 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; Coronary Artery Disease; Cancer; Chronic Kidney Diseases; COPD; Obesity; Sickle Cell Disease; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease; Neoplasms; Renal Insufficiency, Chronic; Pulmonary Disease, Chronic Obstructive; Obesity; Anemia, Sickle Cell; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Eligible patients who don't opt out will be randomized to one of two arms (automated call vs text messaging)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated call (Active Comparator): Patients receive up to two automated phone calls in English or Spanish depending the patients' language indicated in their electronic health record (EHR), between the hours of 10:00am and 9:00pm Monday through Friday.
  Interventions: Other: Community outreach method
- Text messaging (Active Comparator): Patients receive up to two text messages in English or Spanish depending the patients' language indicated in their electronic health record (EHR), between the hours of 10:00am and 9:00pm Monday through Friday.
  Interventions: Other: Community outreach method

INTERVENTIONS:
Other: Community outreach method — The method includes automated call and text messaging to increase testing for COVID-19

SUMMARY:
As part of National Institutes of Health Rapid Acceleration of Diagnostics-Underserved Populations (RADx-UP) program, the goal of the RADxUP study is to develop, test, and evaluate a rapid, scalable capacity building project to enhance COVID-19 testing in three regional community health centers (CHCs) in San Diego County, California. In collaboration with CHC partners, their consortium organization, Health Quality Partners (HQP), investigators are pursuing the following Specific Aims: 1) Compare the effectiveness of automated calls vs text messaging for uptake of COVID-19 testing among asymptomatic adult patients with select medical conditions and those 65 years of age and older receiving care at participating CHCs. Secondarily, investigators will invite all study participants to receive flu vaccination and will assess feasibility and acceptability of study participants to refer adult family household members who are essential workers for COVID-19 testing. 2) Gather patient, provider, CHC leadership, and community stakeholder insights to establish best practices for future scale-up of COVID-19 testing sustainability and vaccination.

DETAILED DESCRIPTION:
Pronounced inequities and disparities in coronavirus disease (COVID-19)COVID-19 morbidity and mortality have been reported, largely due to comorbid conditions and social determinants of health. Approximately 95% of COVID-19 related deaths occur among individuals with underlying medical conditions. Of all racial/ethnic groups, Hispanic/Latino communities in San Diego County have experienced the greatest burden of COVID-19 disease and deaths. Furthermore, testing challenges to date are evident, including long turnaround of test results and longer waiting times for African American and Hispanics compared to whites. The goal of this community-engaged proposal is to develop, test, and evaluate a rapid, scalable capacity building project to enhance COVID-19 testing in three regional community health centers (CHCs) in San Diego County. In collaboration with CHC partners, their consortium organization (Health Quality Partners), and community stakeholders, investigators propose the following Specific Aims: 1) Compare the effectiveness of automated and live prompts and reminders and their combination for uptake of COVID-19 testing among adult patients with select medical conditions or those 65 years of age and older receiving care at participating CHCs. Secondarily, investigators will invite all study participants to receive flu vaccination and will assess feasibility and acceptability of study participants to refer adult family household members who are essential workers for COVID-19 testing. 2) Gather patient, provider, CHC leadership, and community stakeholder insights to establish best practices for future scale-up of COVID-19 testing sustainability and vaccination. This community-engaged project includes underserved (socioeconomically disadvantaged and large proportion of Hispanic/Latinos) as well as COVID-19 vulnerable individuals (patients with medical comorbidities and 65 years of age and older). The approach considers regional COVID-19 morbidity and mortality disparities to identify strategies to address disproportionate infection rates and follow-up. By working in partnership with health care providers, health care system leaders, and community stakeholders, the research team has the potential to build the evidence-base approaches and identify sustainable solutions to understand and address the current and future pandemics in underserved and vulnerable populations.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will include asymptomatic men and women receiving care at participating community health centers with at least one clinic visit in the last year, age 21 years and over, with co-morbid conditions deemed by the Centers for Disease Control and Prevention to increase risk for severe COVID-19 illness, including heart failure, coronary artery disease, cancer, chronic kidney diseases, COPD, obesity, sickle cell disease and type 2 diabetes mellitus, and those 65 years of age and older.

Exclusion Criteria:

* Under age 21, inability to communicate in English and other study languages, inability to complete anterior nasal swab sampling for COVID-19

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9120 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Martinez, PhD, Principal Investigator — Moores Cancer Center, University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Community health center staff will mail an introductory letter to eligible individuals describing the importance of COVID-19 testing, inviting them to receive a test, offering opt out instructions, and noting that follow-up contact (phone call, text message) will take place if they do not opt out. Patients who do not opt out and those whose mail is not returned will be randomized one week after the introductory letter is mailed.
Pre-assignment Details: Participants will be randomized to one of two arms: test messaging and automated call
Period: Overall Study
Arm/Group | Automated Call | Text Messaging
Started | 4489 | 4631
Completed | 12 | 25
Not Completed | 4477 | 4606
Not completed — Lost to Follow-up | 4477 | 4606

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Automated Call | Text Messaging | Total
Number analyzed (Participants) | 12 | 25 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (13) | 57 (13) | 61 (13)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participants has missing value for demographic variables.
  Participants
    number analyzed (Participants) | 12 | 24 | 36
    Female | 8 | 11 | 19
    Male | 4 | 13 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One participants has missing value for demographic variables.
  Participants
    number analyzed (Participants) | 12 | 24 | 36
    Asian | 2 | 1 | 3
    Non-Hispanic White | 2 | 3 | 5
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Hispanic | 7 | 20 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Tested Patients
Description: The percentage of patients who undergo testing within one month of initial contact (automated call vs text messaging) and by the end of the study period (to consider individuals who could not come to the clinic within one month)
Time Frame: 1 month
Population: Because of extremely low testing uptake, slow accrual at participating health centers and continuously changing COVID pandemic, our team was forced to terminate the intervention study and pivot to alternate strategies. Because the study was terminated, the data of the percentage of patients who undergo testing by the end of the study period (automated call vs text messaging) was not collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Automated Call | Text Messaging
Number analyzed (Participants) | 4489 | 4631
Participants | 12 | 25

2. Primary Outcome: Number (%) Tested (Total and by Clinic)
Description: Number (%) of patients who complete COVID-19 test (total and by clinic)
Time Frame: 1 month
Population: Because of extremely low testing uptake, slow accrual at participating health centers and continuously changing COVID pandemic, we were forced to terminate the intervention study and pivot to alternate strategies. This would allow us to continue our efforts to deliver as many COVID-19 tests as possible to help limit the spread of COVID-19 in underserved communities. Because of extremely low participants, there was no power to conduct statistical analysis for primary and secondary outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Automated Call | Text Messaging
Number analyzed (Participants) | 4489 | 4631
Participants | 12 | 25

3. Primary Outcome: Number (%) Infected (Total and by Clinic)
Description: Number (%) of patients with positive COVID-19 test (total and by clinic)
Time Frame: 1 month
Population: Because of extremely low testing uptake, slow accrual at participating health centers and continuously changing COVID pandemic, our team was forced to terminate the intervention study and pivot to alternate strategies. This would allow us to continue our efforts to deliver as many COVID-19 tests as possible to help limit the spread of COVID-19 in underserved communities.
Measure: Count of Participants; unit: Participants
Arm/Group | Automated Call | Text Messaging
Number analyzed (Participants) | 12 | 25
Participants | 0 | 0

4. Primary Outcome: Timeliness of Testing
Description: From time of contact to testing
Time Frame: 1 month
Population: Because of extremely low testing uptake, slow accrual at participating health centers and continuously changing COVID pandemic, our team was forced to terminate the intervention study and pivot to alternate strategies. This would allow us to continue our efforts to deliver as many COVID-19 tests as possible to help limit the spread of COVID-19 in underserved communities. Because the study was terminated, the data of timeliness from time of contact to testing was not collected.
Arm/Group | Automated Call | Text Messaging
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number Vaccinated With Flu Vaccine
Description: Number of patients who receive flu vaccine
Time Frame: 1 month
Population: Because of extremely low testing uptake, slow accrual at participating health centers and continuously changing COVID pandemic, we were forced to terminate the intervention study and pivot to alternate strategies. Because of extremely small number of participants, there was no power to conduct statistical analysis for both primary and secondary outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Automated Call | Text Messaging
Number analyzed (Participants) | 12 | 25
Participants | 9 | 21

6. Secondary Outcome: Proportion of Patients Who Refer for Testing
Description: The proportion of study participants with eligible household members who refer household member(s) for COVID-19 testing
Time Frame: 1 month
Population: Because of extremely low testing uptake, slow accrual at participating health centers and continuously changing COVID pandemic, we were forced to terminate the intervention study and pivot to alternate strategies. This would allow us to continue our efforts to deliver as many COVID-19 tests as possible to help limit the spread of COVID-19 in underserved communities. Because the study was terminated, this data was not collected.
Arm/Group | Automated Call | Text Messaging
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Household Members Referred for Testing
Description: The number of household members referred for COVID-19 testing
Time Frame: 1 month
Population: as for outcome 6
Arm/Group | Automated Call | Text Messaging
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Because of extremely low testing uptake, slow accrual at participating health centers and continuously changing COVID pandemic, our team was forced to terminate the intervention study and pivot to alternate strategies. Because the study was terminated with extremely small number of participants, the adverse events were not monitored/assessed,
Description: Because of extremely low testing uptake, slow accrual at participating health centers and continuously changing COVID pandemic, our team was forced to terminate the intervention study and pivot to alternate strategies. Because the study was terminated with extremely small number of participants, the adverse events were not monitored/assessed,
Arm/Group | Automated Call | Text Messaging
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Because of extremely low testing uptake, slow accrual at participating health centers and continuously changing COVID pandemic, our team was forced to terminate the intervention study and pivot to alternate strategies. This would allow us to continue our efforts to deliver as many COVID-19 tests as possible to help limit the spread of COVID-19 in underserved communities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT05315908/Prot_SAP_000.pdf